CLINICAL TRIAL: NCT06833866
Title: Phase I Trial of 5-Fluorouracil (5FU) -Based Therapy in Combination With Hydroxytyrosol (HT) in Patients With Advanced or Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Maen Abdelrahim, MD, PhD, Pharm.B, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00038031
Record Dates: First submitted 2025-01-15; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Advanced or Metastatic CRC
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 3,4-dihydroxyphenylethanol; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hydroxytyrosol (HT) in combination with Folfiri/Folfox (Experimental): Patients will receive: 1 capsule of HT 25 mg daily for 2 weeks before beginning 5FU-based therapy (FOLFIRI/FOLFOX + Biologics), 1 capsule of HT (25 mg) daily for 2 weeks while receiving the FOLFIRI/FOLFOX + Biologics, until sign of disease progression.
  The prescribed FOLFIRI/FOLFOX administer as: Irinotecan 180 mg/m² intravenously (IV) over 90 minutes concurrently with Leucovorin 400 mg/m² IV over 120 minutes, followed by Fluorouracil 400-500 mg/m² IV bolus then 2400-3000 mg/m² IV infusion over 4-6 hours with or without, the designated Biologics, a standard dose of Cetuximab or Bevacizumab will be administered in 2-week cycles until disease progression or un-tolerated toxicity
  Interventions: Drug: Hydroxytyrosol

INTERVENTIONS:
Drug: Hydroxytyrosol — Patients will receive: 1 capsule of HT 25 mg daily for 2 weeks before beginning 5FU-based therapy (FOLFIRI/FOLFOX + Biologics), 1 capsule of HT (25 mg) daily for 2 weeks while receiving the FOLFIRI/FOLFOX + Biologics, until sign of disease progression.
  The prescribed FOLFIRI/FOLFOX administer as: Irinotecan 180 mg/m² intravenously (IV) over 90 minutes concurrently with Leucovorin 400 mg/m² IV over 120 minutes, followed by Fluorouracil 400-500 mg/m² IV bolus then 2400-3000 mg/m² IV infusion over 4-6 hours with or without, the designated Biologics, a standard dose of Cetuximab or Bevacizumab will be administered in 2-week cycles until disease progression or un-tolerated toxicity
  Other Names: Folfiri/Folfox

SUMMARY:
This is a phase I study investigating the safety and antitumor activity of 5FU-based therapy (FOLFIRI/FOLFOX + Biologics) in combination with Hydroxytyrosol (HT) as a treatment for patients with advanced or metastatic colorectal cancer.

Patients will receive: 1 capsule of HT 25 mg daily for 2 weeks before beginning 5FU-based therapy (FOLFIRI/FOLFOX + Biologics), 1 capsule of HT (25 mg) daily for 2 weeks while receiving the FOLFIRI/FOLFOX + Biologics, until sign of disease progression.

The prescribed FOLFIRI/FOLFOX administer as: Irinotecan 180 mg/m² intravenously (IV) over 90 minutes concurrently with Leucovorin 400 mg/m² IV over 120 minutes, followed by Fluorouracil 400-500 mg/m² IV bolus then 2400-3000 mg/m² IV infusion over 4-6 hours with or without, the designated Biologics, a standard dose of Cetuximab or Bevacizumab will be administered in 2-week cycles until disease progression or un-tolerated toxicity

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all the following criteria are met:

1. Male or female ≥18 years of age.
2. Histopathologically or cytologically confirmed advanced or metastatic CRC.
3. Patient who is eligible for first-line therapy for advanced or metastatic CRC, such as 5FU-based therapy.
4. Measurable disease per the RECIST v1.1.
5. Eastern Cooperative Oncology Group performance status of 0 or 1.
6. Life expectancy ≥6 months.
7. Females of childbearing potential must agree to use birth control during the study and for 30 days after your last dose of HT, at least 9 months after your last dose of oxaliplatin, at least 3 months after your last dose of 5-FU, and at least 6 months after your last dose of irinotecan.
8. Male who are sexually active and their partner can become pregnant, must agree to use birth control during the study and for 30 days after their last dose of HT, at least 6 months after their last dose of oxaliplatin, at least 3 months after his last dose of 5-FU, and at least 3 months after his last dose of irinotecan.

   -

Exclusion Criteria:

Subjects must meet all the inclusion criteria listed above in Section 10.1 and none of the following exclusion criteria:

1. Hematology laboratory values of:

   1. WBC of <3000 and absolute neutrophil count ≤1500 cells/mm3 with the Fy null phenotype.
   2. Platelets ≤100,000 cells/mm3
   3. Hemoglobin ≤9 g/dL (Fe infusion is allowed to correct anemia in iron deficient anemia patients, per standard-of-care)
2. Hepatic laboratory values of aspartate transaminase or alanine aminotransferase:

   1. >5 × upper limits of normal (ULN) if the documented history of hepatic metastases; or
   2. >2.5 × ULN if no liver metastases are present.
3. Serum albumin <2.8 g/dL.
4. Total bilirubin >1.5 × ULN or >1.5 mg/dL.
5. Prothrombin time (PT) or international normalized ratio (INR) >1.5 × ULN. Note: Patients receiving therapeutic doses of anticoagulant therapy may be considered eligible if PT and INR are within the acceptable institutional therapeutic limits.
6. Estimated glomerular filtration rate <50 mL/min.
7. Positive pregnancy test, pregnant, or breastfeeding (female patients only).
8. Any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study.
9. Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study including, but not limited to:

   1. Arrhythmia
   2. Bradycardia
   3. Tachycardia
   4. Symptomatic valvular disease
   5. Symptomatic congestive heart failure classified by the New York Heart Association as Class III or IV
   6. Unstable angina pectoris.
10. Myocardial infarction within the past 6 months.
11. Active bleeding diathesis (platelets less than 100,000 or active bleeding)
12. Current complaints of persistent constipation or history of chronic constipation, bowel obstruction, or fecaloma within the past 6 months.
13. Receiving chronic treatment with corticosteroids ≥5 mg of prednisone per day (or equivalent) or other immunosuppressive agents
14. Known history and/or uncontrolled hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV)-1 or HIV-2.
15. History of galactose intolerance, deficiency of Lapp lactase, or glucose-galactose malabsorption.
16. Receipt of live, attenuated vaccine (e.g., intranasal influenza, measles, mumps, rubella, varicella) or close contact with someone who has received a live, attenuated vaccine within the past 1 month. Note: Influenza vaccine will be allowed if administered >21 days.
17. Receipt of any investigational agent or study treatment within the past 30 days.
18. Receipt of any protein or antibody-based therapeutic agents (e.g., growth hormones or monoclonal antibodies) within the past 3 months.
19. Patients must be able to swallow oral capsules.
20. Participants with metastatic CRC and microsatellite instability-high or deficient mismatch repair tumors.
21. surgical Surgery, within 12-months or less.
22. For patients to be treated with bevacizumab: history of gastrointestinal fistula or perforation, major surgery within 28 days of study treatment initiation, recent hemorrhage, arterial thromboembolic events or deep venous thrombosis within 6 months, uncontrolled hypertension (i.e., BP > 150/90 mm Hg), proteinuria, and hemoptysis.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety, Toxicity, and Pharmacokinetic/Pharmacodynamic (PK/PD) Profile of HT in Combination with FOLFIRI/FOLFOX + Biologics | Through study completion, up to 2 years
  Evaluation of safety profile, toxicity, and PK/PD parameters in patients receiving HT with 5FU-based therapy according to NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) at 6 and 12 Months | 6 and 12 months post study drug initiation
  Measurement of PFS at 6 months and 12 months, based on tumor assessment using RECIST v1.1 criteria.
Objective Response Rate (ORR) According to RECIST v1.1 | Through study completion, up to 2 years
  Proportion of patients achieving partial response (PR) or complete response (CR) as per RECIST v1.1.

OTHER OUTCOMES:
Changes in Health-Related Quality of Life (QoL) | Baseline, 6 months, and 12 months
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).
Immune T-Cell Profiling in Blood and Tissue Samples | Baseline, 2 weeks after HT initiation, and up to 100 weeks (from baseline to disease progression)
  Analysis of T-cell clusters in pretreatment tissue and blood and on-treatment blood (after 2 weeks on HT alone).
  Evaluation of CD4+, CD8+ T cells, and CD8+ T-cell:Treg ratio using multiplexed IF & single-cell RNA sequencing (scRNA-seq).
Assessment of Tissue Immune Cells | Baseline and post-treatment biopsy (up to 100 weeks, at disease progression or prior to surgery, if applicable)
  Quantification of tissue immune cells using flow cytometry.
Analysis of Regulatory Proteins and Plasma Cytokines | Baseline and post-treatment biopsy (up to 100 weeks, at disease progression or prior to surgery, if applicable)
  Evaluation of regulatory proteins and plasma cytokines using a multiplexed protein array.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Esmail, MD, Study Director — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist., Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided